CLINICAL TRIAL: NCT00925522
Title: Clinical Evaluation of Therapy Cool Path Duo Cardiac Ablation System for the Treatment of Ischemic Ventricular Tachycardia (VT)
Brief Title: Therapy Cool Path Ablate VT
Acronym: Ablate-VT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study data no longer needed
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G080076
Record Dates: First submitted 2009-06-08; First posted 2009-06-22 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Ischemic Ventricular Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapy Cool Path Duo Cardiac Ablation System (Experimental): All patients who are eligible receive cardiac ablation procedure for Ischemic Ventricular Tachycardia
  Interventions: Device: Therapy Cool Path Duo Cardiac Ablation System

INTERVENTIONS:
Device: Therapy Cool Path Duo Cardiac Ablation System — Cardiac Ablation Procedure for Ischemic VT using a flexible, insulated 7F all braided catheter that contains an internal lumen connected to 12 open conduits at the 4mm tip electrode for infusion of heparinized saline during radiofrequency ablation; records intracardiac electrograms and can be utilized for cardiac simulation during diagnostic electrophysiologic studies/evaluation.
  1500T9-VT generator is a microprocessor-controlled device that produces a continuous unmodulated radiofrequency (RF) output of 485 kHz. The Generator will be used in Temperature Control mode only. The catheter delivers the RF power from the generator in a monopolar mode between its distal electrode (tip electrode) and a large indifferent electrode.

SUMMARY:
To demonstrate that ablation with the Therapy Cool Path Duo cardiac ablation system can eliminate ischemic VT and that its use does not result in an unacceptable risk of serious adverse events.

DETAILED DESCRIPTION:
Ventricular Tachycardia (VT) is a common complication of ischemic heart disease that is often life threatening. Ventricular tachycardia is defined as three or more beats of ventricular origin in succession at a rate greater than 100 beats per minute. There are no normal QRS complexes associated with VT, and the rhythm is usually regular. Patients with VT experience unpleasant heart palpitations, dyspnea, and syncope, all of which decrease their overall quality of life. They also suffer the consequences of impaired hemodynamics, loss of cardiac efficiency, and are at an increased risk of sudden cardiac death (SCD), which accounts for approximately half of all deaths from patients with cardiovascular disease.

Historically, antiarrhythmic medications served as the first line therapy for the treatment of VT, in spite of low efficacy and high recurrence rates. But in recent years, internal cardioverter defibrillators (ICDs) have become the treatment of choice. Although, ICDs are effective in terminating most arrhythmias, rarely does so without some episodes requiring poorly tolerated shock therapy. Ablative therapy offers an important option for frequent control with the potential for long-term VT elimination. Radiofrequency catheter ablation offers the ability to provide immediate control of recurrent VT. Since the early 2000's, strategies, tools, and techniques have been improving to identify key ablation sites and to deliver effective lesions.

Radiofrequency ablation is successful in treating some but not all arrhythmias. With non irrigated technology it has been difficult to ablate ischemic VT. This may be due to an inadequate lesion size. Irrigated electrodes were developed to create larger lesions. Open irrigation at the catheter tip not only produces larger lesions, but also helps reduce the risk of coagulum (clots) and charring due to high temperatures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has an ICD (Implantable Cardiac Defibrillator) or will be implanted with one prior to discharge of ablation procedure
* Patient has had at least 2 documented spontaneous episode of sustained ischemic VT (Ventricular Tachycardia) within the previous 6 months
* Patient is resistant, intolerant or refractory to at least one Class I or III AAD (Anti-Arrhythmic Drug)
* Patient has been informed of the nature of the study and has agreed to its provisions and provided written informed consent approved by the Institutional Review Board

Exclusion Criteria:

* Non-ischemic VT
* History of stroke or transient ischemic attack within 6 months prior to enrollment
* MI or previous cardiac surgery within 2 months prior to enrollment
* Patient is pregnant or nursing
* Patient has chronic NYHA (New York Heart Association) class IV heart failure
* Limited life expectancy of 6 months or less
* Patient is currently participating in another investigational drug or device study
* Patient is unable or unwilling to cooperate with the study procedures
* Known presence of intracardiac thrombi
* Severe aortic stenosis or flailed mitral valve
* Major contraindication to anticoagulation therapy or coagulation disorder
* Left Ventricular Ejection Fraction <10%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Neal Kay, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Loyola University Medical Center, Maywood, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with atrial flutter are evaluated by ablation doctor in the EP clinic and assessed for possibility of meeting other inclusion criteria.
Pre-assignment Details: This is a non-randomized study.
Groups:
- Therapy Cool Path Duo Cardiac Ablation System: Therapy Cool Path Duo Cardiac Ablation System: Consists of following three system components:
  A flexible, insulated 7F all braided catheter that contains an internal lumen connected to 12 open conduits at the 4mm tip electrode for infusion of heparinized saline during radiofrequency ablation; records intracardiac electrograms and can be utilized for cardiac simulation during diagnostic electrophysiologic studies/evaluation.
  The 1500T9-VT generator is a microprocessor-controlled device that produces a continuous unmodulated radiofrequency (RF) output of 485 kHz. The Generator will be used in Temperature Control mode only. The catheter delivers the RF power from the generator in a monopolar mode between its distal electrode (tip electrode) and a large indifferent electrode.
  The Cool Point ™ Irrigation Pump and Cool Point™ Tubing Set is an external volumetric pump that is intended for use in administration of general I.V. fluids to patient's vascular system through the cat
Period: Overall Study
Arm/Group | Therapy Cool Path Duo Cardiac Ablation System
Started | 20
Completed | 0
Not Completed | 20
Not completed — study closed -- business decision | 20

BASELINE CHARACTERISTICS:
Groups:
- Therapy Cool Path Duo Cardiac Ablation System: Therapy Cool Path Duo Cardiac Ablation System: Consists three system components:
  A flexible, insulated 7F all braided catheter that contains an internal lumen connected to 12 open conduits at the 4mm tip electrode for infusion of heparinized saline during radiofrequency ablation; records intracardiac electrograms and can be utilized for cardiac simulation during diagnostic electrophysiologic studies/evaluation.
  The 1500T9-VT generator is a microprocessor-controlled device that produces a continuous unmodulated radiofrequency (RF) output of 485 kHz. The Generator will be used in Temperature Control mode only. The catheter delivers the RF power from the generator in a monopolar mode between its distal electrode (tip electrode) and a large indifferent electrode.
  The Cool Point ™ Irrigation Pump and Cool Point™ Tubing Set is an external volumetric pump that is intended for use in administration of general I.V. fluids.
Arm/Group | Therapy Cool Path Duo Cardiac Ablation System
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety is Defined as the Incidence of Intra-procedural, Acute or Sub-chronic, Serious Cardiac Adverse Events, up to 7 Days Post-procedure.
Time Frame: 7 days
Measure: Number; unit: participants
Groups:
- Therapy Cool Path Duo Catheter: All patients received RF (radio frequency) therapy from ablation catheter.
Arm/Group | Therapy Cool Path Duo Catheter
Number analyzed (Participants) | 20
participants | 7

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition of AEs and SAEs per clinicaltrials.gov were used
Groups:
- Therapy Cool Path Duo Cardiac Ablation System: Therapy Cool Path Duo Cardiac Ablation System: Consists of:
  A flexible, insulated 7F all braided catheter that contains an internal lumen connected to 12 open conduits at the 4mm tip electrode for infusion of heparinized saline during radiofrequency ablation; records intracardiac electrograms and can be utilized for cardiac simulation during diagnostic electrophysiologic studies/evaluation.
  The 1500T9-VT generator is a microprocessor-controlled device that produces a continuous unmodulated radiofrequency (RF) output of 485 kHz. The Generator will be used in Temperature Control mode only. The catheter delivers the RF power from the generator in a monopolar mode between its distal electrode (tip electrode) and a large indifferent electrode.
  The Cool Point ™ Irrigation Pump and Cool Point™ Tubing Set is an external volumetric pump that is intended for use in administration of general I.V. fluids to patient's vascular system through the catheter in the hospital environment.
Arm/Group | Therapy Cool Path Duo Cardiac Ablation System
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy Cool Path Duo Cardiac Ablation System (N=20)
Arrhythmia(s) including AFL, AF or VT (Cardiac disorders) | 5 (5)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Cardiac Effusion without Tamponade (Cardiac disorders) | 1 (1)
Cardiac Effusion with Tamponade (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapy Cool Path Duo Cardiac Ablation System (N=20)
Hypotension (Cardiac disorders) | 3 (3)
Hypertension (Cardiac disorders) | 3 (3)
Arrythmia (Cardiac disorders) | 2 (2)
Infection (Blood and lymphatic system disorders) | 1 (1)
Chest Pains Palpitations (Cardiac disorders) | 2 (3)
Anxiety/Depression (Psychiatric disorders) | 1 (1)
CHF symptoms (Cardiac disorders) | 2 (3)
Sleep Apnea (Nervous system disorders) | 1 (1)
Hyperlipidemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval from St. Jude Medical prior to any publication.